CLINICAL TRIAL: NCT00719225
Title: Belatacept for Renal Allograft Recipients: A Compassionate Use Program
Brief Title: A Belatacept Compassionate Use Study for Patients With a Kidney Transplant
Status: No longer available | Type: Expanded Access
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: IM103-056
Record Dates: First submitted 2008-07-17; First posted 2008-07-21 (Estimated); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Renal Transplantation
MeSH Terms: interventions — Abatacept

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: Belatacept — IV, 5 mg/kg, once monthly, until BMS terminates trial or Belatacept is available commercially
  Other Names: LEA29Y; BMS-224818

SUMMARY:
To make belatacept available for recipients of a renal allograft who are currently intolerant to or have contraindications to CNIs and/or m-TOR inhibitors and are either:

* unable to construct an adequate immunosuppression regimen due to nonrenal toxicity / contraindication (and withdrawing the causative agent would lead to renal graft loss) OR
* at imminent risk of losing the allograft kidney due to nephrotoxicity and have no other options for renal replacement therapy

ELIGIBILITY:
Please call 800-398-9157 for information on this study

Inclusion Criteria:

* Men and women of age 18 years or older inclusive
* Recipient of a renal allograft for at least ≥ 2 months
* EBV positive
* Unable to tolerate a suitable immunosuppression regimen to prevent acute allograft rejection, due to:
* Extra-renal toxicity related to CNIs and/or m-TOR inhibitors that is refractory to medical management (eg, uncontrolled seizures)
* Contraindication to CNIs and/or m-TOR inhibitors

OR

* At imminent risk of losing allograft kidney due to nephrotoxicity
* Renal failure: ≥ Stage 4 on KDOQI Scale (GFR 15 - 29 cc/min)
* And no other renal replacement therapy
* Subjects must be receiving the maintenance immunosuppressants MMF, MPA, or AZA

Exclusion Criteria:

* Any significant infection, extra-renal solid organ (heart, liver, pancreas) or cell (islet, bone marrow, stem cell) transplants, with an unresolved episode of AR within the last 6 weeks
* EBV negative

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (7):
- United States (7):
  - Scripps Green Hospital, La Jolla, California
  - Office Of Dr. Allan Kirk, Atlanta, Georgia
  - Acadiana Renal Physicians, New Iberia, Louisiana
  - Tulane Abdominal Transplant Institute, New Orleans, Louisiana
  - UNC Kidney Center, Chapel Hill, North Carolina
  - The Transplant Center Of The Lehigh Valley, Allentown, Pennsylvania
  - Texas Transplant Physician'S Group, San Antonio, Texas

REFERENCES:
- See also: EAP Investigator Requests — https://www.bms.com/healthcare-providers/early-patient-access-to-investigational-medicine/investigational-drugs-available.html
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm